CLINICAL TRIAL: NCT07140302
Title: Stereotactic Surgical Management of Dystonia: Efficacy and Safety
Brief Title: Surgery of Dystonia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Mostafa, assistant lecture, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25-8-1MD
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Dystonia Stereotactic Surgery
MeSH Terms: interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stereotactic surgery of dystonia (Experimental): Patients with dystonia undergoing stereotactic surgical management (either Deep Brain Stimulation or Radiofrequency Lesioning), with choice of procedure determined by clinical indication.
  Interventions: Procedure: deep brain stimulation

INTERVENTIONS:
Procedure: deep brain stimulation — Stereotactic implantation of DBS electrodes with chronic electrical stimulation of target nuclei for dystonia.
  or Stereotactic radiofrequency ablation of dystonia-related target nuclei.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and clinical outcomes of stereotactic surgery (Deep Brain Stimulation or Radiofrequency Lesioning) in patients with dystonia.

The main questions it aims to answer are:

* Does stereotactic surgery improve dystonia severity as measured by the Burke-Fahn-Marsden Dystonia Rating Scale - Motor (BFMDRS-M)?
* Are the procedures safe, with an acceptable complication profile during follow-up?

Participants will:

* Undergo stereotactic surgery for dystonia (either Deep Brain Stimulation or Radiofrequency Lesioning, based on clinical indication).
* Be followed postoperatively for assessment of motor function and adverse events at the first postoperative week and six months after surgery.

DETAILED DESCRIPTION:
Detailed Description

Dystonia is a chronic movement disorder characterized by sustained or intermittent muscle contractions, resulting in abnormal postures, repetitive movements, and functional disability. Medical therapy often provides limited benefit, particularly in patients with severe or refractory forms of dystonia.

Stereotactic surgical approaches, including Deep Brain Stimulation (DBS) and Radiofrequency (RF) lesioning, have emerged as effective treatment options for carefully selected patients. DBS offers a reversible and adjustable method of neuromodulation, while RF lesioning provides a less resource-intensive option in settings where DBS may not be feasible.

The purpose of this study is to evaluate the clinical outcomes and safety of stereotactic surgical management in patients with dystonia treated at our center. All enrolled participants will undergo stereotactic surgery-either DBS implantation or RF lesioning-based on clinical indications and multidisciplinary decision-making.

Patients will be assessed preoperatively and followed postoperatively at standardized intervals, including the first postoperative week and at six months. The primary outcome is the change in dystonia severity as measured by the Burke-Fahn-Marsden Dystonia Rating Scale - Motor Subscale (BFMDRS-M). Secondary outcomes will include functional disability, quality of life, and perioperative complications.

This study is designed as a prospective interventional case series without a formal control group, aiming to provide real-world outcome data on the effectiveness and safety of stereotactic surgical management of dystonia

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with dystonia with at least 1-year duration since symptom onset.
* Inadequate relief of dystonia following treatment with standard pharmacotherapies (e.g., levodopa, clonazepam, trihexyphenidyl, or baclofen) or botulinum toxin injections.

Exclusion Criteria:

* Previous DBS surgery.
* Underwent DBS combined with another surgical procedure for dystonia (e.g., lesioning or peripheral denervation).
* Cognitive dysfunction or other neuropsychiatric disorders.
* Progressive neurological conditions other than dystonia.
* Coagulopathy or bleeding disorders.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in Dystonia Severity (BFMDRS-Motor Score) | From baseline (within 4 weeks prior to surgery) to the first postoperative week and up to 6 months postoperatively.
  Change in motor severity of dystonia as assessed by the Burke-Fahn-Marsden Dystonia Rating Scale - Motor Subscale (BFMDRS-M; range 0-120, higher scores = worse dystonia). The primary endpoint is the percent change from baseline to follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Faculity of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
may be shared